CLINICAL TRIAL: NCT06223178
Title: Efficacy of Thumb-tack Needle Treatment for Diminished Ovarian Reserve: Study Protocol for a Randomized Controlled Trial
Brief Title: Efficacy of Thumb-tack Needle Treatment for Diminished Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaomei Shao (Other)
Collaborators: Hangzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023ZX010-DOR
Record Dates: First submitted 2023-12-20; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Diminished Ovarian Reserve
Keywords: Diminished Ovarian Reserve; Acupoint; Thumb-tack Needle; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thumb-tack needle acupuncture (Experimental): 53 Patients in this group will achieve 24 sessions treatment of thumb-tack needle in 12 consecutive weeks. Treatment will be operated by trained acupuncturists.
  Interventions: Device: thumb-tack needle; Other: Basic gynecological treatment
- Sham acupuncture group (Sham Comparator): A sham thumb-tack needle, which has no difference in appearance with the verum thumb-tack needle but is lack of needle, are used for 53 patient in this group. 24 sessions of treatment will be performed in 12 consecutive weeks. Treatment will be operated by trained acupuncturists.
  Interventions: Device: sham thumb-tack needle; Other: Basic gynecological treatment

INTERVENTIONS:
Device: thumb-tack needle — Sterilizing skin and avoiding vessels, the thumb-tack needle are directly stock to the surface of acupoints by a band-aid, kneading and pressing for 5 minutes. The thumb-tack needle will be embedded in the skin and keep staying for 72 hours. Patients will be taught to press them 3 to 4 times per day. As tolerated by them, each pressing will lasts 1 minutes with an interval of about 4 hours.
  Arms: Thumb-tack needle acupuncture
Device: sham thumb-tack needle — Sterilizing skin and avoiding vessels, the sham thumb-tack needle are directly stock to the surface of acupoints by a band-aid, kneading and pressing for 5 minutes. The sham device will be embedded in the skin and keep staying for 72 hours. Patients will be taught to press them 3 to 4 times per day. As tolerated by them, each pressing will lasts 1 minutes with an interval of about 4 hours.
  Arms: Sham acupuncture group
Other: Basic gynecological treatment — Gynecological health care guidance will be provided as patients needed.

SUMMARY:
Diminished Ovarian Reserve (DOR) is characterized as an important cause of infertility. Acupuncture has been extensively used to treat female infertility. This study was conducted to investigate the efficacy of thumb-tack needle，as a new special type of acupuncture and long-lasting treatment modality,in the treatment of DOR.

DETAILED DESCRIPTION:
There will be a multi-center, randomized, sham-controlled trial. 106 patients will be randomly assigned into thumb-tack needle acupuncture or sham-acupuncture in 1:1 ratio. All the patents will achieve 12 sessions of verum or sham treatments in 20 weeks(12 weeks for treatment and 8 weeks for follow-up). Patients, outcome assessors and statisticians are masked from group assignment. The study is aim to evaluate the efficacy of thumb-tack needle for DOR.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age < 40 years old, female;
* Clinical diagnosis of Diminished Ovarian Reserve: meet both items in twice tests with an interval of at least 4 weeks(tested between 2rd to 4th day of menstrual cycle):

  1. 10 IU/L < FSH < 20 IU/L,
  2. Anti-Müllerian hormone(AMH) < 1.1ng/mL.
* without any mind disease, willing to participate in the study and sign the informed consent.
* without any other treatment.

Exclusion Criteria:

* Low or no response to exogenous gonadotropins, or with congenital anomalies in the development of the reproductive tract；
* Pregnant or breastfeeding;
* Abnormal body temperatures at the moment;
* Psychopath, alcoholic, Patient with severe depression, history of substance abuse and severe primary diseases of cardiovascular, liver, kidney and hematopoietic system;
* Currently enrolled in other clinical trials or refuse to cooperate with the study protocol.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
changes of serum follicle-stimulating hormone (FSH) level | baseline，week 4, week 12，week 20(week 8 in follow-up)
  The increasing of serum follicle-stimulating hormone（FSH） is one of the main symptoms of Diminished Ovarian Reserve. The normal value of FSH is 1.37-9.9 U/L in follicular phase, and higher the FSH value, the worse ovarian function. Patients in this study will be asked to take the serum FSH text between day2 to day4 of menstrual period in whole observation. Patients with amenorrhea take every 28 days as a supposed menstrual cycle instead.

SECONDARY OUTCOMES:
changes of 1.Serum Anti-Müllerian Hormone (AMH) level | baseline，week 12, week 20(week 8 in follow-up)
  AMH is another recommend index to measure ovarian function. Compared to FSH, Anti-Müllerian Hormone has less fluctuation and more accuracy. The normal value of serum AMH is 2-6.8ng/ml in follicular phase, and lower the value, the worse condition.
temperature of sensitized acupoint | baseline，week 4, week 12，week 20(week 8 in follow-up)
  "Acupoint sensitization" suggests that there are specific changes of biological characteristics on the body surface or acupuncture points in a pathological state. Acupoints associated with the disease may manifest as sensitivity to pain and heat. Infrared thermography (IRT) will be used to measured the temperature of the DOR-related acupoints.
pain threshold of sensitized acupoint | baseline，week 4, week 12，week 20(week 8 in follow-up)
  Pain threshold of DOR-related acupoints will be tested by pressure pain threshold gauge (PTG).
the modified Kupperman Index(KI) | baseline，week 4, week 12，week 20(week 8 in follow-up)
  The modified Kupperman Index (KI) is widely used for female self-evaluation of the severity of menopausal symptoms in clinical practice. It values 13 items of menopausal symptoms on a scale of 0 to 3. The final score of KI is the sum of each score multiplied with the base score respectively, ranging from 0-63. The final KI score is less than 6 means normal, between 6 to 15 are classified as mild, 16 to 30 as moderate, and greater than 30 as severe.
Self-Rating Anxiety Scale (SAS) | baseline，week 4, week 12，week 20(week 8 in follow-up)
  According to the frequency of symptom occurrence, the SAS contains 20 items reflecting subjective feelings of anxiety, and each item is rated on a four-point scale of 1 to 4, including 15 positive and 5 negative items. 1 means never, 2 is for sometimes, 3 is for frequently, 4 is always. Positive items are rating from 1-4, while negative items is from 4 to 1. Once the evaluation is complete, the scores for each of the 20 items are added together as score X. Score X will multiply by 1.25 and then round to the nearest whole number to obtain a standardized score Y, which is the final result of SAS. According to the Chinese normative results, the cut-off value of the SAS standardized score is 50, where 50-59 is mild anxiety, 60-69 is moderate anxiety, and 69 or more is severe anxiety.
Self-rating Depression Scale (SDS) | baseline，week 4, week 12，week 20(week 8 in follow-up)
  The SDS also contains 20 items reflecting subjective feelings of depression, with 10 positive and 10 negative ratings. 1 means never, 2 is for sometimes, 3 is for frequently, 4 is always. Positive items are rating from 1-4, while negative items is from 4 to 1. Once the evaluation is complete, the scores for each of the 20 items are added together as score X. Score X will multiply by 1.25 and then round to the nearest whole number to obtain a standardized score Y, which is the final result of SDS.The cut-off value of SDS standardized score is 53, where 53 to 62 is considered as mild depression, 63 to 72 is moderate depression, and 72 or more is severe depression.
Psychological constitution of traditional Chinese medicine(TCM） | baseline，week 4, week 12，week 20(week 8 in follow-up)
  The TCM psychological constitution scale is compiled by Professor Wang Qi of Beijing University of Chinese Medicine, which is widely used in clinical practice. There are 9 items and 66 small items in the TCM constitution scale, and it requires patients fill the scale truthfully by themselves according to their real situation in the last year. Nine psychological constitutions will be determined by conversion score: mild constitution, qi deficiency constitution, qi depression constitution, yin deficiency constitution, yang deficiency constitution, blood stasis constitution, special constitution, phlegm-dampness constitution and damp-heat constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hangzhou, Zhejiang, China